CLINICAL TRIAL: NCT05278195
Title: Assessing the Prognosis of Transarterial Chemoembolization in Combination With PD-1/PD-L1 Inhibitors and Molecular Target Therapies(VEGF-TKI/Bevacizumab) for Hepatocellular Carcinoma by Using Clinical and Imaging Biomarkers
Brief Title: Assessing the Prognosis of TACE in Combination With PD-1/PD-L1 Inhibitors and Molecular Target Therapies for HCC by Using Clinical and Imaging Biomarkers
Acronym: CHANCEsub
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Other Study IDs: CHANCE-Biomarker
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; immune checkpoint iInhibitors; transarterial chemoembolization; real-world study
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to id

transarterial chemoembolization (TACE) in combination with immune checkpoint inhibitors (ICIs) and molecular targeted therapies in patients with hepatocellular carcinoma (HCC) .

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
2. Has not received any previous systemic therapy for HCC (including chemotherapy, molecularly targeted therapy, immunotherapy);
3. Both PD-1/PD-L1 inhibitors and anti-angiogenesis drugs patients received only include marketed drugs but are not limited to HCC approval;
4. TACE was performed up to 3 months after the first PD-1/PD-L1 inhibitor/anti-angiogenic drug treatment or within 1 month before treatment;
5. Received at least 1 cycle of PD-1/PD-L1 inhibitor/anti-angiogenic drug combination therapy after TACE treatment；

7. Has repeated measurable intrahepatic lesions according to RECIST v1.1;

Exclusion Criteria:

1. Cholangiocarcinoma, fibrolamellar, sarcomatoid hepatocellular carcinoma, and mixed hepatocellular/cholangiocarcinoma subtypes(confirmed by histology, or pathology) are not eligible;
2. Unable to meet criteria of combination timeframe described above;
3. Missing follow-up data;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate HCC who received TACE in combination with PD-1/PD-L1 inhibitors and molecular target therapies under real-world practice conditions.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death due to any cause.

SECONDARY OUTCOMES:
Specificity | baseline
  The specificity of the radiomics artificial intelligence model for identifying optimal candidates among patients who treated TACE in combination with PD-1/PD-L1 inhibitors and molecular target therapy will be calculated.
Sensitivity | baseline
  The sensitivity of the radiomics artificial intelligence model for identifying optimal candidates among patients who treated TACE in combination with PD-1/PD-L1 inhibitors and molecular target therapy will be calculated.
The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of the radiomics artificial intelligence mode | baseline
  The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of the radiomics artificial intelligence model for identifying optimal candidates among patients who treated TACE in combination with PD-1/PD-L1 inhibitors and molecular target therapy will be calculated.
Accuracy | baseline
  Defined by a confusion matrix of sensitivity and specificity to true positives and true negatives.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, M.D., Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llovet JM, Villanueva A, Marrero JA, Schwartz M, Meyer T, Galle PR, Lencioni R, Greten TF, Kudo M, Mandrekar SJ, Zhu AX, Finn RS, Roberts LR; AASLD Panel of Experts on Trial Design in HCC. Trial Design and Endpoints in Hepatocellular Carcinoma: AASLD Consensus Conference. Hepatology. 2021 Jan;73 Suppl 1:158-191. doi: 10.1002/hep.31327. Epub 2020 Sep 9. No abstract available. PMID 32430997
- [Background] Llovet JM, Kelley RK, Villanueva A, Singal AG, Pikarsky E, Roayaie S, Lencioni R, Koike K, Zucman-Rossi J, Finn RS. Hepatocellular carcinoma. Nat Rev Dis Primers. 2021 Jan 21;7(1):6. doi: 10.1038/s41572-020-00240-3. PMID 33479224
- [Background] Ochoa de Olza M, Navarro Rodrigo B, Zimmermann S, Coukos G. Turning up the heat on non-immunoreactive tumours: opportunities for clinical development. Lancet Oncol. 2020 Sep;21(9):e419-e430. doi: 10.1016/S1470-2045(20)30234-5. PMID 32888471
- [Background] Pinato DJ, Murray SM, Forner A, Kaneko T, Fessas P, Toniutto P, Minguez B, Cacciato V, Avellini C, Diaz A, Boyton RJ, Altmann DM, Goldin RD, Akarca AU, Marafioti T, Mauri FA, Casagrande E, Grillo F, Giannini E, Bhoori S, Mazzaferro V. Trans-arterial chemoembolization as a loco-regional inducer of immunogenic cell death in hepatocellular carcinoma: implications for immunotherapy. J Immunother Cancer. 2021 Sep;9(9):e003311. doi: 10.1136/jitc-2021-003311. PMID 34593621
- [Derived] Jin ZC, Zhou JW, Chen JJ, Ding R, Scheiner B, Wang SN, Li HL, Shen QX, Lu QY, Liu Y, Zhang WH, Luo B, Shi HB, Huang M, Wu YM, Yuan CW, Huang MS, Li JP, Wu JB, Zhu XL, Zhong BY, Zhou HF, Wang YQ, Gu SZ, Peng ZY, Zheng CS, Liu RB, Xu GH, Yang WZ, Xu AB, Liu DF, Qi X, Yeo YH, Zhu HD, Zhao Y, Pinato DJ, Ji F, Teng GJ. Longitudinal Body Composition Identifies Hepatocellular Carcinoma With Cachexia Following Combined Immunotherapy and Target Therapy (CHANCE2213). J Cachexia Sarcopenia Muscle. 2024 Dec;15(6):2705-2716. doi: 10.1002/jcsm.13615. Epub 2024 Nov 27. PMID 39604073